CLINICAL TRIAL: NCT03521167
Title: Multimodal Analgesia Versus Traditional Opiate Based Analgesia and Cardiac Surgery Outcome
Brief Title: Multimodal Analgesia Versus Traditional Opiate Based Analgesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAvsTOBA
Record Dates: First submitted 2018-04-12; First posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Cardiac Surgery
MeSH Terms: interventions — Ketamine; Lidocaine; Dexmedetomidine; Gabapentin; Acetaminophen

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- T (No Intervention): traditional opioid based regimen
- MD (Active Comparator): multimodal group with dexmedetomidine
  Interventions: Drug: Ketamine; Drug: Lidocaine; Drug: Dexmedetomidine; Drug: Gabapentin; Drug: Tylenol; Drug: Gabapentin Pill; Drug: Tylenol Pill
- M (Placebo Comparator): multimodal with saline placebo
  Interventions: Drug: Ketamine; Drug: Lidocaine; Drug: Gabapentin; Drug: Tylenol; Drug: Gabapentin Pill; Drug: Tylenol Pill

INTERVENTIONS:
Drug: Ketamine — Intraoperatively use. 0.5 mg/kg with induction bolus, followed by 5mcg/kg/min infusion after induction.
  Continue up to 1 hour prior to extubation. maximum total dose 3mg/kg.
  Arms: M; MD
Drug: Lidocaine — Intraoperatively use. start lidocaine infusion at 2mg/min after anesthesia induction, and continue up to 1 hour prior to extubation.
  Arms: M; MD
Drug: Dexmedetomidine — Intraoperatively use. start dexmedetomidine infusion at 0.5 mcg/kg/min after anesthesia induction, and continue up to 1 hour prior to extubation.
  Arms: MD
Drug: Gabapentin — Postoperatively use. 300 mg PO TID starting POD1 until discharge Use lower dose for >65y or if patient having significant sedation/dizziness
  Arms: M; MD
Drug: Tylenol — Postoperatively use. 1000 mg PO Q8hr starting POD0 until discharge (max 3000 mg in 24hrs) Reduce to 650 mg PO Q6h if <70kg
  Arms: M; MD
Drug: Gabapentin Pill — Pre-operatively use. 300mg PO up to 1 hour before OR time Reduce to 100 mg PO in patients >65y or with GFR < 50 Consider dose reduction in patients with sleep apnea
  Arms: M; MD
Drug: Tylenol Pill — Pre-operatively use. 1000 mg PO up to 1 hour before OR time Reduce to 650 mg PO if <70kg Don't use if h/o liver disease or anticipated liver injury (right heart failure, pulmonary hypertension, etc leading to systemic venous congestion)
  Arms: M; MD

SUMMARY:
Pain after cardiac surgery can be moderate to severe with incisions to the sternum and lower extremities, and also the placement of chest tubes. Postoperative pain may contribute to delirium, stress, myocardial oxygen demand supply imbalance, etc. Traditionally postoperative pain management after cardiac surgery has been based on opiate analgesics. However, opiates have many deleterious side effects including nausea/vomiting, ileus, bladder dysfunction, and respiratory depression, which substantially influence patient recovery and may delay discharge after surgery.

The current study is designed to evaluate if an opiate sparing multimodal regimen of tylenol, gabapentin, ketamine, lidocaine and dexmedetomidine provided better analgesic effect (pain score, postoperative PCA opioid dose), less side effects (PONV) and improved cardiac surgery outcome (delirium, a-fib, AKI, dysglycemia) compared to a traditional fentanyl and hydromorphine regimen after cardiac surgery. Additionally, it aims to investigate if the benefit of multimodal regimen is achieved by combination of all drugs or all drugs except dexmedetomodine by introducing third group of study patients who will be randomized to all interventions except saline placebo instead of dexmedetomodine infusion.

ELIGIBILITY:
Inclusion Criteria:

* ASA II-III Grade
* BMI 18-31kg/m2
* Adult patients presenting for on-pump cardiac surgery through median sternotomy

Exclusion Criteria:

* Cardiac surgery without sternotomy
* emergency surgery
* h/o allergy to any of the medications in the research protocol
* hepatic disease with elevated liver enzymes (preoperative SGPT and SGOT elevated to 1.5 times maximum normal value)
* pregnancy
* unable to give consent
* preoperative mental disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of analgesic effect | Within 3 months after surgery
  Evaluation of analgesic effect by Visual Analogue Scale

SECONDARY OUTCOMES:
Additional opioid consumption | Within 3 days after operation
  assessed by daily sufentanil PCIA dose
postoperative delirium | Within 3 days after operation
  evaluated by CAM-ICU criteria

CONTACTS AND LOCATIONS:
Overall Officials: Lin Jin, PHD, Principal Investigator — Fudan University